CLINICAL TRIAL: NCT05619523
Title: An Intervention to Promote Positive Peer Relationships and Reduce Prejudice and Bias in Childhood
Brief Title: Developing Inclusive Youth: Promoting Intergroup Friendships and Inclusive Classrooms in Childhood
Acronym: DIY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Melanie Killen, Professor of Human Development and Quantitative Methodology, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Developing Inclusive Youth; 5R01HD093698-04 (NIH)
Record Dates: First submitted 2022-10-27; First posted 2022-11-17 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Social Exclusion; Prejudice, Racial; Prejudice; Sexism; Peer Group
Keywords: intergroup attitudes; prejudice; bias; sexism; racism; exclusion; classroom intervention; moral reasoning; intergroup friendships; child development
MeSH Terms: conditions — Social Isolation; Racism; Prejudice; Sexism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: DIY Tool Classrooms (Experimental): Developing Inclusive Youth (DIY) classrooms complete a pretest and posttest survey in addition to completing 8 scenarios using the DIY online tool and a class discussion for each scenario.
  Interventions: Behavioral: Developing Inclusive Youth (DIY)
- Control: Business As Usual Classrooms (No Intervention): The control group follows a Business-As-Usual plan (no "alternative" program is implemented for the control group.) They complete a pretest and posttest in the same weeks as the experimental group.

INTERVENTIONS:
Behavioral: Developing Inclusive Youth (DIY) — Developing Inclusive Youth (DIY) is a web-based curriculum tool that serves as the intervention program. The animated and narrated tool displays eight peer social exclusion scenarios in a range of familiar everyday social contexts (such as the playground and school). Children enter their responses while watching the scenarios. Responses include making decisions about inclusion and exclusion, evaluating the actions as okay or not okay, attributing feelings to includers, excluders, and excluded characters, and selecting reasons that best match their justification for their decisions and evaluations. The program includes teacher-guided group discussions following use of the tool in which teachers facilitate discussions about children's interpretations of the scenarios, evaluations, reflections regarding their own experiences of exclusion, and solutions. Participants will view and discuss 8 scenarios and engage in a discussion for each one over the course of 8 weeks.
  Other Names: Developing Inclusive Youth; DIY
  Arms: Intervention: DIY Tool Classrooms

SUMMARY:
The goal of this clinical trial is to test the beneficial impacts of a web based intervention program called Developing Inclusive Youth for children in 3rd, 4th, and 5th grade. The main questions it aims to answer are:

* Does the Developing Inclusive Youth (DIY) program, which is a web-based curriculum tool with a teacher-led classroom discussion, reduce prejudicial attitudes and biases as well as increase intergroup friendships for a sample of 8 -11 year old children enrolled in 3rd , 4th, and 5th grade U.S. classrooms?
* Does the Developing Inclusive Youth (DIY) program lead to grade-related, gender-related and ethnic-related differences regarding reducing prejudicial attitudes and increasing intergroup friendships?
* Does the Developing Inclusive Youth (DIY) program change teacher attitudes regarding the malleability of prejudice, the importance of intergroup friendships, and comfort levels with discussing social inclusion and exclusion experiences in the classroom?

Student participants will take 15-20 minutes to use a Chrome notebook and headphones to access the online tool and the teacher will then lead a classroom discussion lasting 25-30 minutes. The intervention program will occur once a week for eight weeks.

The student outcome measures, given at pretest and posttest, are also assessed with Chrome notebooks while children are sitting at their desks in the classroom. The outcome measures take 25-30 minutes. Researchers will compare children in the intervention classes to children in other classes of the same grade at their school to see if the tool promotes positive peer relationships and reduces prejudice and bias.

Teacher participants will take a 25-minute online pretest and posttest survey in their classroom to assess their theories of prejudice, their awareness of their students' intergroup friendships, comfort with discussing peer social inclusion and exclusion in class, and their awareness of student experiences of exclusion.

DETAILED DESCRIPTION:
A within school randomized control trial intervention design will be implemented to promote intergroup relationships and reduce prejudice in childhood for children between 7 and 12 years of age, enrolled in grades 3, 4, and 5 in U.S. elementary public schools. The intervention students watch an online tool for 15 minutes accompanied by a 30-minute teacher-led classroom discussion. Students in the control condition will be business as usual. There will be 720 students and 36 teachers, reflecting an ethnically diverse population. The outcome measures assess school belonging, peer and teacher classroom support, trait attributions of diverse peers, social evaluations about intergroup exclusion as well as the likelihood of exclusion, and math and science competency beliefs of diverse peers. All teachers participate in a 2-hour training session prior to the start of the school semester. All participating students have active parental consent. All teachers take a survey about their theories of prejudice, awareness of student experiences with exclusion, and strategies for talking about peer conflict in the classroom prior to the beginning of the program and provide their assent. There is high fidelity of the program due to the delivery of the information which is online. There are many steps in place to ensure fidelity of the teacher component which involves leading the classroom discussion. Multi-level analyses will be employed to determine whether the students in the intervention improve in their desire for intergroup friendships and experiences of classroom support relative to the students in the control condition. Novel data will be collected regarding intergroup attitudes held by children across a range of target groups and grade levels. The information from this project is expected to improve peer relationships due to the more positive classroom environment and an increase of social inclusion among peers. All children are expected to benefit by their participation in the program with a goal of improving academic engagement and healthy child development.

ELIGIBILITY:
For Child Participants

Inclusion Criteria:

* children with parental consent in grades 3, 4, or 5 at participating schools
* be between the ages of 7 and 12 years
* children who need assistance sitting at their desk or reading the text can participate provided that an adult mentor is assigned to them to assist with the protocol

For Teacher Participants:

* teachers of students in grades 3, 4, and 5 at participating schools and who provide assent
* no age limits for teacher participation

Exclusion Criteria:

* school has identified the student as unable to participate due to disability status.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 885 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Montgomery, Study Chair — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodenow, C. (1993). The psychological sense of school membership among adolescents: Scale development and educational correlates. Psychology in the Schools, 30, 79-90. DOI:10.1002/1520-6807.
- [Background] Van Ryzin MJ, Gravely AA, Roseth CJ. Autonomy, belongingness, and engagement in school as contributors to adolescent psychological well-being. J Youth Adolesc. 2009 Jan;38(1):1-12. doi: 10.1007/s10964-007-9257-4. Epub 2007 Nov 30. PMID 19636787
- [Background] Collie, R. J., Martin, A. J., Papworth, B. & Gins, P., (2016). Students' interpersonal relationships, personal best (PB) goals, and academic engagement, Learning and Individual Differences, 45, 65-76. http://dx.doi.org/10.1016/j.lindif.2015.12.002
- [Background] Liben LS, Bigler RS. The developmental course of gender differentiation: conceptualizing, measuring, and evaluating constructs and pathways. Monogr Soc Res Child Dev. 2002;67(2):i-viii, 1-147; discussion 148-83. PMID 12465575
- [Background] Mulvey KL, Rizzo MT, Killen M. Challenging gender stereotypes: Theory of mind and peer group dynamics. Dev Sci. 2016 Nov;19(6):999-1010. doi: 10.1111/desc.12345. Epub 2015 Sep 22. PMID 26395753
- [Background] Bierman, K. L., & McCauley, E. (1987). Children's descriptions of their peer interactions: Useful information for clinical child assessment. Journal of Clinical Child Psychology, 16(1), 9-18. https://doi.org/10.1207/s15374424jccp1601_2
- [Background] Grutter J, Gasser L, Zuffiano A, Meyer B. Promoting Inclusion Via Cross-Group Friendship: The Mediating Role of Change in Trust and Sympathy. Child Dev. 2018 Jul;89(4):e414-e430. doi: 10.1111/cdev.12883. Epub 2017 Jun 19. PMID 28626994
- [Background] Killen M, Burkholder AR, D'Esterre AP, Sims RN, Glidden J, Yee KM, Luken Raz KV, Elenbaas L, Rizzo MT, Woodward B, Samuelson A, Sweet TM, Stapleton LM. Testing the effectiveness of the Developing Inclusive Youth program: A multisite randomized control trial. Child Dev. 2022 May;93(3):732-750. doi: 10.1111/cdev.13785. Epub 2022 May 25. PMID 35612354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited elementary schools in the local public school district by sending an email invitation to every school in the district. Once the schools elected to participate, families received hard copy or electronic consent forms in English, Spanish, and/or Mandarin. Students who returned consent forms received an eraser. Participating schools received $1500 and teachers with students in the intervention group received $150 to compensate for their time administering the program.
Pre-assignment Details: Teachers were potential participants who were screened for the purpose of determining eligibility, but who did not participate and thus were not considered enrolled, due to the low frequency of potential participants (N = 51). Teachers whose students were in the intervention group were compensated for giving up instructional time to the intervention and for helping facilitate delivery of the program.
Period: Overall Study
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Started | 522 | 363
Completed | 522 | 363
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms | Total
Number analyzed (Participants) | 522 | 363 | 885
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 522 | 363 | 885
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.67 (.95) | 9.72 (1.01) | 9.69 (.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 180 | 431
  Male | 271 | 183 | 454
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 74 | 59 | 133
  Black | 62 | 42 | 104
  Latine | 74 | 45 | 119
  Multiracial | 68 | 59 | 127
  White | 191 | 122 | 313
  Other/Unknown | 53 | 36 | 89
Region of Enrollment [Number; unit: participants]
  United States | 522 | 363 | 885

OUTCOME MEASURES:

1. Primary Outcome: School Belonging Scale
Description: The School Belonging Scale is an 8-item self-report measure consisting of a rating scale ranging from 1 (really not true) to 6 (really true). The average of all items creates a final score of perceived school belonging in which higher scores indicate higher levels of perceived school belonging. The original Psychological Sense of School Membership scale (PSSM) (Goodenow, 1999) measure has been found to have internal consistency reliability for both suburban (0.875) and urban (0.803) elementary school populations. We modified this measure for length. Pilot testing revealed that this new, shorter version was also found to have high internal reliability (0.714). The construct validity of the scale was also indicated through a significant relationship with teacher-ratings of student social standing (Goodenow, 1993).
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 4.72 (.07) | 4.72 (.09)

2. Primary Outcome: Classroom Life Scale: Peer Personal Support Subscale Personal Support Subscale
Description: This is a five-item measure including items about whether other students in my class care about me and other students in my class like me for who I am. The measure has been found to produce reliability figures of .92 (Van Ryzin, Gravely, & Roseth, 2009) and our modified version utilizing a 6-point response scale in place of the original 5-point scale found similar reliability scores (0.896). The rating scale ranged from 1 (really not true) to 6 (really true). The average of all items creates a score of perceived peer personal support in which higher scores indicate higher levels of perceived peer support. Performance on the Van Ryzin et al. (2009) scale has been demonstrated to have an independent positive effect on engagement in learning and has been validated by connections to academic engagement (Collie, Martin, Papworth, and Gins, 2016).
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 4.35 (.08) | 4.40 (.11)

3. Primary Outcome: Classroom Life Scale: Teacher Personal Support Subscale
Description: The degree to which students perceive their teachers as personally supportive will be assessed using this 4-item measure. Items include statements such as my teacher cares about me and my teacher likes me for who I am. This measure was also modified from the original rating scale to a 6-point rating scale, which ranged from 1 (really not true) to 6 (really true). Van Ryzin et al. (2009) reported an internal consistency reliability of .91, and our pilot testing found a similar internal consistency reliability, 0.893.
  A composite score was computed using the mean of all items in the scale. Scores ranged from a minimum of 1 to a maximum of 6. A higher score indicated higher teacher support, the more desirable outcome.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 5.12 (.06) | 5.03 (.09)

4. Primary Outcome: Trait Attributions for Gender, Race, & Ethnicity
Description: An adaptation of the Child Occupations and Traits (COAT) scale (Liben & Bigler, 2002; 0.99) measures stereotypes re: gender and race intergroup categories. Participants respond to three types of items (e.g., how smart or not smart; how hardworking or lazy; or friendly or mean) and this measure was also modified to utilize a 6 point rating scale. There are two sub-categories, gender and race. The questions probe the degree to which children assign traits to specific groups. The version we utilized contained 12 items, 6 about race and 6 about gender and pilot testing revealed that this version had a high internal reliability for the full scale (0.919), as well as for the gender and the race subcomponents (0.859 and 0.849, respectively).
  Scores ranged from a minimum of 1 to a maximum of 6. A higher score indicates more positive (better) trait attributions about peers.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 502 | 343
score on a scale | 4.83 [4.45 to 5.36] | 4.82 [4.39 to 5.25]

5. Primary Outcome: High Status Occupation Expectations
Description: This set of items is adapted from Liben & Bigler (2002). These items probe participant perceptions of the likelihood of group members obtaining high status occupations. Participants were asked "Which kid do you think will grow up to be a [pilot/doctor/lawyer/scientist]?" with one item for each profession. Participants selected which child of 8 possible choices they thought would become the profession. The 8 choices included a boy and a girl of each of the following racial groups: Asian, Black, Latine, White. The measure was made binary by whether participants selected an underrepresented minority (URM) (Black or Latine) in high status professions, or whether they selected a race group that is not underrepresented (White or Asian). The goal of the intervention was that more students in the treatment condition selected a URM student after the intervention program. Therefore in the fields below, the category Underrepresented Minority (URM) indicates the number of participants who select
Time Frame: one week following completion of the 8-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 499 | 342
Participants
  Doctor: Underrepresented Minority (URM) | 204 | 131
  Doctor: Highly represented group (non-URM) | 295 | 211
  Lawyer: Underrepresented Minority (URM) | 269 | 185
  Lawyer: Highly represented group (non-URM) | 230 | 157
  Pilot: Underrepresented Minority (URM) | 215 | 143
  Pilot: Highly represented group (non-URM) | 284 | 199
  Scientist: Underrepresented Minority (URM) | 185 | 138
  Scientist: Highly represented group (non-URM) | 314 | 204

6. Primary Outcome: Reported Contact Scale
Description: The diversity of friendships will be assessed using an adaptation of the Friendship Questionnaire (Bierman & McCauley, 1987). The original measure has been widely utilized to assess the quality and quantity of children's peer interactions and has proven to be reliable (ranges from .72 to .82). The adaptation consisted of adding the intergroup categories of gender and race/ethnicity. This adapted version was also found to be internally reliable (0.659). Using gender, racial, and ethnic background, we will record how often they play with outgroup peers to determine the proportion of cross-gender, cross-race, and cross-ethnic playmate interactions.
  Scores on the scale ranged from a minimum of 1 to a maximum of 6. Higher scores indicate a higher level of reported cross-group contact, which is the more desirable outcome.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 3.34 [3.00 to 3.67] | 3.31 [3.00 to 3.67]

7. Primary Outcome: Desire for Intergroup Contact
Description: This assessment consists of 5 separate items about how much the child wants to play with X, where X refers to pictures of girls, boys, and kids who are depicted as African American, European American, and Asian American). Response choices are provided on a 6 point rating scale ranging from 1 (really do not want to) to 6 (really want to). During pilot testing this measure was found to have a high internal consistency reliability (0.767). Using students' gender, ethnic, and racial background, we will record their desire to play with outgroup peers to determine the proportion of cross-gender, cross-race and cross-ethnic playmate preferences.
  Scores on the scale ranged from a minimum of 1 to a maximum of 6. Higher scores indicate a higher desire for intergroup contact, the more desirable outcome.
Time Frame: change, one week following completion of the 8-week intervention
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 343
score on a scale | 3.99 [3.33 to 4.67] | 3.92 [3.17 to 4.58]

8. Primary Outcome: Personal Experiences With Exclusion
Description: This assessments consists of 8 items about whether the child experiences exclusion in a school context. Response choices are provided on a 5 point Likert-type rating scale ranging from "Never" to "Always." This measure has been validated in previous research (Killen et al., 2022).
  Scores on the scale range from a minimum score of 1 and maximum score of 5. Higher scores indicate higher levels of personal experiences of exclusion, which is the less desirable outcome. Thus the goal of the intervention is to result in lower scores in the treatment group at posttest.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 2.02 (.06) | 1.96 (.08)

9. Primary Outcome: Evaluations of Exclusion in Intergroup and Same Group Contexts
Description: This assessment consists of 2 items repeated 4 times to reflect different race and gender combinations for a total of 8 items. This measure is adapted from Cooley et al., 2019. The items ask participants to evaluate exclusion in an intergroup and same group social context. Responses were on a 6-point Likert-type scale ranging from 1 (really not okay) to 6 (really okay).
  Scores on this scale range from a minimum of 1 to a maximum of 6. A higher score on this scale indicates viewing exclusion as more acceptable and a lower score indicates viewing exclusion as less acceptable. The goal of the intervention is to promote lower scores, indicating participants are less accepting of exclusion.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 3.05 (.07) | 2.96 (.09)

10. Primary Outcome: Likelihood of Inclusion in Intergroup and Same Group Contexts
Description: This assessment consists of 5 items repeated 4 times to reflect different race and gender combinations for a total of 20 items. This measure is adapted from Cooley et al., 2019. The items ask participants to predict the likelihood of a child inviting someone to their birthday party, where the children they can invite may be of the same or a different race. Responses were on a 6-point Likert-type scale ranging from 1 (very unlikely) to 6 (very likely).
  Scores on this scale range from a minimum of 1 to a maximum of 6. Higher scores indicate participants expect intergroup inclusion to be more likely, which is the more desirable outcome.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 4.53 (.05) | 4.54 (.06)

11. Primary Outcome: Stereotypes About Inclusivity
Description: This scale is adapted from Liben and Bigler (2002). The scale probes participant perceptions of the inclusivity levels of different groups. These scales were created consistent with the literature on gender stereotypes (Berenbaum, Martin, & Ruble, 2015; Mulvey, Rizzo, & Killen, 2016). A 5 point rating scale ranging from 1 (none) to 5 (all) indicates the proportion of children within a hypothetical target group whom participants believe fit into a categorization. Pilot testing revealed 0.800 for the 5-item measure of inclusivity levels of different groups.
  Scores on this scale range from a minimum of 1 to a maximum of 5. Higher scores indicate more positive beliefs about peers' inclusive behavior, the more desirable outcome.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 3.70 [3.17 to 4.08] | 3.75 [3.17 to 4.17]

12. Primary Outcome: Stereotypes About Math & Science Competence
Description: This scale is adapted from Liben and Bigler (2002). The scale probes participant perceptions of the math and science abilities of different groups. This scale was created consistent with the literature on gender stereotypes (Berenbaum, Martin, & Ruble, 2015; Mulvey, Rizzo, & Killen, 2016). A 5 point rating scale ranging from 1 (none) to 5 (all) indicates the proportion of children within a hypothetical target group whom participants believe fit into a categorization. Pilot testing revealed 0.796 for the 5-item measure of math and science abilities of different groups.
  Scores ranged from a minimum of 1 and a maximum of 5. Higher scores indicate more positive beliefs about peers' math and science abilities, which is the more desirable outcome.
Time Frame: one week following completion of the 8-week intervention
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
Number analyzed (Participants) | 522 | 363
score on a scale | 4.89 [4.58 to 5.39] | 4.89 [4.50 to 5.25]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Intervention: DIY Tool Classrooms | Control: Business As Usual Classrooms
All-Cause Mortality (participants affected / at risk) | 0/522 | 0/363
Serious Adverse Events (participants affected / at risk) | 0/522 | 0/363
Other Adverse Events (participants affected / at risk) | 0/522 | 0/363

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT05619523/Prot_001.pdf
  • Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT05619523/SAP_002.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT05619523/ICF_000.pdf